CLINICAL TRIAL: NCT05904769
Title: Non-invasive Measurement of Blood Glucose, Blood Pressure and Extrapolation of QRS Complex Using a Wrist Wearable Photoplethysmography Sensor
Brief Title: A Study of Non-invasive Measurement of Blood Glucose and Blood Pressure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of staffing support
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Narayan (Guru) G. Kowlgi, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-010799
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hospitalized Diabetic Group (Experimental): Subjects hospitalized and diabetic on insulin, undergoing four times daily blood sugar checks, will wear the LIFELEAF Smartwatch for the duration of their hospital stay.
  Interventions: Device: LIFELEAF Smartwatch
- Electrophysiologic (EP) Group (Experimental): Subjects undergoing an EP procedure will wear he LIFELEAF Smartwatch for the duration of the procedure.
  Interventions: Device: LIFELEAF Smartwatch

INTERVENTIONS:
Device: LIFELEAF Smartwatch — Noninvasive wearable smartwatch/monitor that utilizes photoplethysmography (PPG) which is a set of measurements acquired from the light flashed from the back of the watch and measuring the intensity of the reflected light from the blood in the blood vessels just below the skin at the wrist. Provides a non-invasive method for measuring blood glucose as well as alternative method for measuring blood pressure, heart rate and rhythm, etc.

SUMMARY:
The purpose of this research is to compare blood glucose, blood pressure and electrocardiogram (ECG) readings on the LIFELEAF Smartwatch compared to standard methods of measurement.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients on insulin undergoing four times daily blood sugar checks as part of standard of care.
* Patients undergoing continuous monitoring for heart rate, ECG and blood pressure as part of their routine care.
* Patients undergoing invasive and noninvasive electrophysiologic procedures.

Exclusion Criteria:

* Patients unable to provide informed consent.
* Patients without arms as these are needed to wear the wrist-based sensor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narayan Guru G. Kowlgi, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Zero subjects were enrolled in the hospitalized diabetic arm as the study was terminated early due to a lack of staffing support.
Groups:
- Hospitalized Diabetic Group: Subjects hospitalized and diabetic on insulin, undergoing four times daily blood sugar checks, wore the LIFELEAF Smartwatch for the duration of their hospital stay.
  LIFELEAF Smartwatch: Noninvasive wearable smartwatch/monitor that utilizes photoplethysmography (PPG) which is a set of measurements acquired from the light flashed from the back of the watch and measuring the intensity of the reflected light from the blood in the blood vessels just below the skin at the wrist. Provides a non-invasive method for measuring blood glucose as well as alternative method for measuring blood pressure, heart rate and rhythm, etc.
- Electrophysiologic (EP) Group: Subjects undergoing an EP procedure wore the LIFELEAF Smartwatch for the duration of the procedure.
  LIFELEAF Smartwatch: Noninvasive wearable smartwatch/monitor that utilizes photoplethysmography (PPG) which is a set of measurements acquired from the light flashed from the back of the watch and measuring the intensity of the reflected light from the blood in the blood vessels just below the skin at the wrist. Provides a non-invasive method for measuring blood glucose as well as alternative method for measuring blood pressure, heart rate and rhythm, etc.
Period: Overall Study
Arm/Group | Hospitalized Diabetic Group | Electrophysiologic (EP) Group
Started | 0 | 87
Completed | 0 | 81
Not Completed | 0 | 6
Not completed — Physician Decision | 0 | 6

BASELINE CHARACTERISTICS:
Population: Zero subjects were enrolled in the hospitalized diabetic arm as the study was terminated early due to a lack of staffing support.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hospitalized Diabetic Group | Electrophysiologic (EP) Group | Total
Number analyzed (Participants) | 0 | 87 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 62.3 (10.24) | 62.3 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 27 | 27
  Male |  | 60 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 87 | 87

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Difference in measurement of Systolic Blood Pressure using the wrist-based PPG sensor versus invasive measurement of blood pressure measured in millimeters of mercury (mmHg).
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hospitalized Diabetic Group | Electrophysiologic (EP) Group
Number analyzed (Participants) | 0 | 81
mmHg |  | 13.08 (17.22)

2. Primary Outcome: Diastolic Blood Pressure
Description: Difference in measurement of Diastolic Blood Pressure using the wrist-based PPG sensor versus invasive measurement of blood pressure measured in millimeters of mercury (mmHg).
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hospitalized Diabetic Group | Electrophysiologic (EP) Group
Number analyzed (Participants) | 0 | 81
mmHg |  | 8.42 (10.56)

3. Primary Outcome: Blood Glucose Level
Description: The difference in measurement of blood glucose levels using the wrist-based PPG sensor versus standard blood-based measurement measured in milligrams per deciliter (mg/dL) in subjects who had standard of care blood glucose monitoring done. Only subjects who are hospitalized and diabetic per standard of care receive standard of care blood-based glucose monitoring.
Time Frame: Baseline
Population: 0 subjects enrolled in the hospitalized diabetic arm as study was terminated early (lack of staffing support). Data not collected for this outcome measure in the EP group as it didn't apply to the EP arm. Standard blood-based glucose measurements were only measured on subjects that were diabetic + hospitalized. EP subjects were not hospitalized; due to this standard blood glucose was not monitored in this group therefore a comparison couldn't be made to the PPG sensor blood glucose measurements.
Groups:
- Electrophysiologic (EP) Group: Subjects undergoing an EP procedure who do not receive daily blood sugar checks wore the LIFELEAF Smartwatch for the duration of the procedure.
  LIFELEAF Smartwatch: Noninvasive wearable smartwatch/monitor that utilizes photoplethysmography (PPG) which is a set of measurements acquired from the light flashed from the back of the watch and measuring the intensity of the reflected light from the blood in the blood vessels just below the skin at the wrist. Provides a non-invasive method for measuring blood glucose as well as alternative method for measuring blood pressure, heart rate and rhythm, etc.
Arm/Group | Hospitalized Diabetic Group | Electrophysiologic (EP) Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through the end of study completion, approximately 24 hours.
Description: Zero subjects were enrolled in the hospitalized diabetic arm as the study was terminated early due to a lack of staffing support.
Arm/Group | Hospitalized Diabetic Group | Electrophysiologic (EP) Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/87
Other Adverse Events (participants affected / at risk) | 0/0 | 0/87

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of staffing support.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT05904769/Prot_SAP_000.pdf